CLINICAL TRIAL: NCT06435663
Title: Fellow Docotor, Master's Degree
Brief Title: The Clinical Application of Ultramicro-flow Technique in the Treatment of Benign Uterine Tumors With High-intensity Focused Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-080
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Patients With Uterine Fibroids Receiving HIFUA Treatment ,and Can Undergo Regular Follow-up

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): In HIFUA treatment, SMI technology was used to evaluate the therapeutic effect. The SMI technology used Toshiba Aplio 800 color ultrasound diagnostic instrument, equipped with SMI imaging software, convex array probe, frequency 1-6 MHz, and color mode ultra fine vessel imaging (eSMI). After the target lesion is determined by abdominal scanning, adjust the depth and gain, and record the number, location, size, shape and boundary of the lesion. CDFI and eSMI models were used to observe the blood supply within the lesion, which were divided into four levels according to Adler grading criteria. Hemodynamic parameters were measured, including peak systolic velocity (PSV) and resistance index (RD). Hemodynamic data were compared to calculate the effectiveness of changes in uterine benign tumor examination after treatment.
  Interventions: Other: Different methods of efficacy evaluation
- control group (Other): In HIFUA treatment, organ ultrasound contrast evaluation technology is used for efficacy evaluation. Sono Vue (Bracco company) is used as the contrast agent. Before use, 5 ml of physiological saline is injected into the bottle, vigorously shaken until the freeze-dried powder is completely dispersed. 1.5 ml of contrast agent is extracted and rapidly injected through the anterior elbow vein, followed by 5 ml of physiological saline injection. After injecting contrast agent, start the timer at the same time, observe under ultrasound imaging, keep the probe stationary during examination, observe continuously for 2 minutes, and store dynamic images. Calculate the effective rate of physical examination changes in benign uterine tumors after treatment by displaying ablation volume through contrast-enhanced ultrasound before and after treatment.
  Interventions: Other: Different methods of efficacy evaluation

INTERVENTIONS:
Other: Different methods of efficacy evaluation — When the treatment method remains unchanged, compare the accuracy data of the effectiveness evaluation between the two groups, and verify that the ultra-fine blood flow imaging technology (SMI) is superior to the organ contrast-enhanced ultrasound evaluation method in the efficacy evaluation after HIFUA treatment.

SUMMARY:
High intensity focused ultrasound ablation (HIFUA) is a new non-invasive treatment method for uterine tumors. Traditionally, nuclear magnetic resonance imaging (NMRI), also known as magnetic resonance imaging (MRI), is used as guidance to focus ultrasound on the fibroid tissue, generating high temperatures of 65-85 ℃, causing protein inactivation, cell apoptosis, and coagulation necrosis of tumor cells. While accurately ablating fibroid tissue, it avoids damaging normal tissue outside the treatment area. Since 2000, a large number of clinical studies have demonstrated the safety and effectiveness of MRI for HIFUA in the treatment of uterine fibroids. In 2013, the Chinese FDA approved MRI guided HIFUA treatment for uterine fibroids. At present, more and more medical institutions in China have introduced this device and carried out non-invasive treatment of uterine fibroids. In March 2020, the Minimally Invasive Treatment Group of the Magnetic Resonance Application Professional Committee of the China Medical Equipment Association designated the "Chinese Expert for MRI Guided Focused Ultrasound Treatment of Uterine Fibroids", making HIFUA more standardized. Superb micro vascular imaging (SMI) is an improved Doppler technology that applies a new adaptive algorithm to remove tissue motion signals and blood flow overflow phenomena, and can clearly display the extremely low velocity blood flow inside the blood vessels. Previous studies have shown that SMI has a significantly higher ability to detect blood vessels in tumors than color Doppler flow imaging (CDFI), and can more sensitively detect the blood flow of microvessels within tumors. This provides a cheap and simple non-invasive examination method for clinical practice, and real-time guidance for treatment can be provided during the treatment process, making it easy to operate and promote in clinical practice.

This study randomly divided all adult patients diagnosed with uterine fibroids or adenomyosis admitted to our hospital from May 2024 to December 2024 into two groups based on the inclusion and exclusion of specimens: 1) Experimental group: HIFUA treatment, treatment efficacy evaluation using SMI technology; control group: HIFUA treatment, treatment efficacy evaluation using organ contrast-enhanced ultrasound technology.

Both groups of subjects need to be followed up: at 3 months, 6 months, and 12 months after treatment, patients will undergo gynecological uterine ultrasound examination at the outpatient department, and the volume of uterine fibroids or adenomyosis will be recorded. The aim of this study is to compare the accuracy data of two groups in evaluating treatment effectiveness, and to verify that ultra-fine blood flow imaging (SMI) technology is superior to organ contrast-enhanced ultrasound in evaluating the efficacy of HIFUA treatment。

DETAILED DESCRIPTION:
Research object All adult patients diagnosed with uterine fibroids or adenomyosis admitted to our hospital from May 2024 to December 2024.

Inclusion criteria Patients with clinically diagnosed uterine fibroids or adenomyosis who meet the following conditions: 1) Imaging shows that the uterine fibroids are located between the muscle walls, or are pedunculated subserosal or submucosal fibroids, which are classified as types 2-6 by the International Federation of Gynecology and Obstetrics (FIGO); The diagnosis of adenomyosis is clear; 2) The imaging shows that there is no intestinal obstruction between uterine fibroids or adenomyosis and the abdominal wall, or the impact of intestinal obstruction can be eliminated through treatment, making it a safe treatment path; 3) Abdominal subcutaneous fat thickness ≤ 4 cm; 4) The farthest distance from the abdominal wall skin to the target area for treating fibroids is ≤ 14 cm; 5) The patient is generally in good condition and can tolerate and maintain a prone position for 2 hours or longer. 6) Adult and infertile women.

Exclusion criteria

1) Unclear clinical diagnosis; 2) Uterine fibroids or adenomyosis rapidly increase in the short term, or imaging suggests a tendency for malignancy, or the malignant potential is uncertain; 3) Acute skin infection in the treatment area; 4) Uncontrolled acute pelvic inflammatory disease; 5) The general condition is poor, with severe dysfunction of important organs such as the heart, liver, and kidneys; 6) Severe coagulation dysfunction; 7) There are large skin scars in the treatment area of the lower abdomen. 8) Sedative and analgesic drugs cannot be used; 9) Postmenopausal enlarged uterine fibroids or adenomyosis. 10) Pregnant women, individuals with mental disorders, cognitive impairments, etc. who are unable to cooperate with treatment.

Materials and Methods Experimental materials

1. Haiying HY2900 ultrasound focusing equipment (Wuxi Haiying Medical Technology Co., Ltd.) Toshiba Aplio i800 color ultrasound diagnostic instrument (Toshiba Medical Systems Co., Ltd.), equipped with SMI imaging software, convex array probe, frequency 1-6MHz, using color mode ultra fine vessel imaging (eSMI);
2. The contrast agent used is sulfur hexafluoride microbubbles for injection (Shanghai Bolaike Xinyi Pharmaceutical Co., Ltd.).

Research methods

Randomly group the included subjects:

1. Experimental group: In HIFUA treatment, SMI technology was used to evaluate the therapeutic effect. The SMI technology used Toshiba Aplio 800 color ultrasound diagnostic instrument, equipped with SMI imaging software, convex array probe, frequency 1-6 MHz, and color mode ultra fine vessel imaging (eSMI). After the target lesion is determined by abdominal scanning, adjust the depth and gain, and record the number, location, size, shape and boundary of the lesion. CDFI and eSMI modes were used to observe the blood supply within the lesion, which were classified into 4 levels according to Adler grading criteria: 0 level, with no blood flow signal inside the fibroid; Grade 1, with a small amount of blood flow signal within the fibroid, with 1-2 short rod-shaped blood flows visible; Level 2, moderate to equal blood flow signal, with one clear blood vessel visible within the fibroid, with a length exceeding the lesion radius or 3-4 short rod-shaped blood flow signals visible; Level 3, rich blood flow, with 4 or more blood vessels visible within the fibroid. The surrounding blood vessels of the fibroid form a network around the entire fibroid, presenting a ball hugging sign, or have multiple branching branches extending into the fibroid, interweaving into a network or patchy pattern. Detect hemodynamic parameters, including peak systolic velocity (PSV) and resistance index (RD), and compare hemodynamic data to calculate the effectiveness of changes in uterine benign tumor physical examination after treatment.
2. Control group: In HIFUA treatment, organ ultrasound contrast evaluation technology was used for efficacy evaluation. Sono Vue (Bracco company) was used as the contrast agent. Before use, 5 ml of physiological saline was injected into the bottle, vigorously shaken until the freeze-dried powder was completely dispersed. 1.5 ml of contrast agent was extracted and rapidly injected through the anterior elbow vein, followed by 5 ml of physiological saline injection. After injecting contrast agent, start the timer at the same time, observe under ultrasound imaging, keep the probe stationary during examination, observe continuously for 2 minutes, and store dynamic images. The CEUS enhancement degree of uterine fibroids can be divided into: high enhancement: the enhancement degree is higher than that of the uterine muscle layer; Equal enhancement: The degree of enhancement is equal to the uterine muscle layer; Low enhancement: The degree of enhancement is lower than that of the uterine muscle layer. Calculate the effective rate of physical examination changes in benign uterine tumors after treatment by displaying ablation volume through contrast-enhanced ultrasound before and after treatment.

Both groups of subjects need to be followed up: at 3 months, 6 months, and 12 months after treatment, patients will undergo gynecological uterine ultrasound examination at the outpatient department, and the volume of uterine fibroids or adenomyosis will be recorded.

Efficacy evaluation: Calculate the volume of uterine fibroids before treatment, ablation rate, and volume reduction rate at 3 months, 6 months, and 12 months. Volume (cm3)=left and right diameter (cm) X anterior and posterior diameter (cm) X long diameter (cm) X 0.523, ablation rate=volume of non perfused area after treatment/volume of uterine fibroids before treatment X 100%, volume reduction rate=(volume of uterine fibroids before treatment - volume of uterine fibroids after 3.6.12 months after treatment)/volume of uterine fibroids before treatment X 100%. Ablation rate of 70% is considered satisfactory, 50% V ablation rate<70% is partial ablation, and ablation rate V 5 (less than 50)% is considered ineffective. SMI evaluates the blood flow signal inside uterine fibroids. Level 0 indicates satisfactory ablation, level 1 indicates partial ablation, and levels 2-3 indicate ineffective ablation 2) Control group: In HIFUA treatment, organ ultrasound contrast evaluation technology was used for efficacy evaluation. Sono Vue (Bracco company) was used as the contrast agent. Before use, 5 ml of physiological saline was injected into the bottle, vigorously shaken until the freeze-dried powder was completely dispersed. 1.5 ml of contrast agent was extracted and rapidly injected through the anterior elbow vein, followed by 5 ml of physiological saline injection. After injecting contrast agent, start the timer at the same time, observe under ultrasound imaging, keep the probe stationary during examination, observe continuously for 2 minutes, and store dynamic images. The CEUS enhancement degree of uterine fibroids can be divided into: high enhancement: the enhancement degree is higher than that of the uterine muscle layer; Equal enhancement: The degree of enhancement is equal to the uterine muscle layer; Low enhancement: The degree of enhancement is lower than that of the uterine muscle layer. Calculate the effective rate of physical examination changes in benign uterine tumors after treatment by displaying ablation volume through contrast-enhanced ultrasound before and after treatment.

Both groups of subjects need to be followed up: at 3 months, 6 months, and 12 months after treatment, patients will undergo gynecological uterine ultrasound examination at the outpatient department, and the volume of uterine fibroids or adenomyosis will be recorded.

Efficacy evaluation: Calculate the volume of uterine fibroids before treatment, ablation rate, and volume reduction rate at 3 months, 6 months, and 12 months. Volume (cm3)=left and right diameter (cm) X anterior and posterior diameter (cm) X long diameter (cm) X 0.523, ablation rate=volume of non perfused area after treatment/volume of uterine fibroids before treatment X 100%, volume reduction rate=(volume of uterine fibroids before treatment - volume of uterine fibroids after 3.6.12 months after treatment)/volume of uterine fibroids before treatment X 100%. Ablation rate of 70% is considered satisfactory, 50% V ablation rate<70% is partial ablation, and ablation rate V 5 (less than 50)% is considered ineffective. SMI evaluates the blood flow signal inside uterine fibroids. Level 0 indicates satisfactory ablation, level 1 indicates partial ablation, and levels 2-3 indicate ineffective ablation

ELIGIBILITY:
Inclusion Criteria:Patients with clinically diagnosed uterine fibroids or adenomyosis who meet the following conditions: 1) Imaging shows that the uterine fibroids are located between the muscle walls, or are pedunculated subserosal or submucosal fibroids, which are classified as types 2-6 by the International Federation of Gynecology and Obstetrics (FIGO); The diagnosis of adenomyosis is clear; 2) The imaging shows that there is no intestinal obstruction between uterine fibroids or adenomyosis and the abdominal wall, or the impact of intestinal obstruction can be eliminated through treatment, making it a safe treatment path; 3) Abdominal subcutaneous fat thickness ≤ 4 cm; 4) The farthest distance from the abdominal wall skin to the target area for treating fibroids is ≤ 14 cm; 5) The patient is generally in good condition and can tolerate and maintain a prone position for 2 hours or longer. 6) Adult and infertile women.Exclusion criteria：1) Unclear clinical diagnosis; 2) Uterine fibroids or adenomyosis rapidly increase in the short term, or imaging suggests a tendency for malignancy, or the malignant potential is uncertain; 3) Acute skin infection in the treatment area; 4) Uncontrolled acute pelvic inflammatory disease; 5) The general condition is poor, with severe dysfunction of important organs such as the heart, liver, and kidneys; 6) Severe coagulation dysfunction; 7) There are large skin scars in the treatment area of the lower abdomen. 8) Sedative and analgesic drugs cannot be used; 9) Postmenopausal enlarged uterine fibroids or adenomyosis. 10) Pregnant women, individuals with mental disorders, cognitive impairments, etc. who are unable to cooperate with treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness | At 3 months, 6 months, and 12 months after treatment
  Record two sets of data on the uterus at 3 months, 6 months, and 12 months after treatment. Size of fibroids, record effective rate data, compare effective rate data between two groups, and compare differences between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No